CLINICAL TRIAL: NCT03910426
Title: Prognostic Determinants (Nutritional Versus Functional Versus Biochemical) of Survival and Quality of Life in Prevalent End-stage Kidney Disease Patients Treated With Dialysis
Brief Title: Prognostic Determinants of Survival and Quality of Life in Prevalent End-stage Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: UGent_EQ5D
Record Dates: First submitted 2019-04-01; First posted 2019-04-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Dialysis; Quality of Life; Nutrition
MeSH Terms: interventions — Blood Specimen Collection; Sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of blood, stool and nails
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling — Blood is sampled before a midweek dialysis session once every year with a maximum of 3 samples in total.
Other: Nails collection — At the occasion of the blood sampling, finger nails are cut and collected.
Other: Stool collection — At the occasion of the blood sampling, patients are asked to bring a stool sample.
Other: Physical Functioning — A subgroup of patients are asked to perform some physical tests.
Other: Sleep — A subgroup of patients are asked to sleep 2-3 nights with a Motionwatch (Actigraphy) to recording their arm movements.

SUMMARY:
Patients with end-stage kidney disease are treated with dialysis to increase their life expectancy as well as their quality of life (QoL). Scientific researchers are currently still looking for markers to evaluate dialysis in an objective way. It has been proven before that the currently clinically used parameters (like the dialysis adequacy parameter Kt/V) are not appropriate enough to estimate dialysis dose.

The current project aims at identifying potential (predicting) biomarkers based on functional capacity, nutritional status and/or QoL.

DETAILED DESCRIPTION:
This multisite study is an observational study during which prevalent dialysis patients are followed during maximum 3 years, and they undergo different tests.

Once a year (max 3 times), blood is sampled, stool is collected, and finger nails are taken all before a midweek session. Demographic data are registered and Davies-Stokes scores are calculated. Blood is analysed for different solutes: e.g. total and free fractions of protein-bound toxins, sedimentation, erythrocytes, hematocrit, leukocytes, thrombocytes, Ferritin, VitB12, Fasting glucose, c-reactive protein, urea, creatinine, albumin, total protein, cholesterol, triglycerides, bilirubin,...

At the same occasion, patients are questioned about different items (QoL, nutrition) by a (study) nurse or coordinator, using different questionnaires: Euroqol 5 dimension scale (EQ-5D), Patient-Reported Outcomes Measurement Information System (Promis-29), and Mini Nutritional Assessment (MNA).

A subgroup of patients were asked to perform some functional tests: Tinetti-Test, Sit to Stand (5 times), Frailty and Injuries: Cooperative Studies on Intervention Techniques (Ficsit) test, 2 or 6 minutes walking test, handgrip strength and quadriceps power measurement, back scratch test, compensatory stepping correction-backward test and skin fold measurement. All tests are non-invasive and are validated for routine measurements in the elderly.

In order to quantify sleep, patients were asked to wear a Motionwatch (Actigraphy) to register their arm movements during 2 or 3 nights as well as to fill out 2 questionnaires related to sleep: Pittsburgh Sleep Quality Index (PSQI) and Insomnia Severity Index (ISI). To compare sleep in dialysis patients with healthy persons, age and gender matched healthy volunteers were also included in the study and were asked to sleep 2 or 3 nights with the Motionwatch and to complete the ISI and PSQI.

Patients who were transplanted got an extra blood sampling just before transplantation as well as 4 months after transplantation.

ELIGIBILITY:
Inclusion Criteria:

- end-stage kidney disease patients treated with dialysis (peritoneal dialysis or hemodialysis)

Exclusion Criteria:

* active inflammation
* malignancy
* cognitive disorder
* not understanding the dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients treated with dialysis were eligible for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between protein-bound uremic toxin concentrations and physical parameter 6 minute walking test (6MWT) | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. As physical parameters, the 6MWT (m) is performed.
Correlation between protein-bound uremic toxin concentrations and physical parameter sit-to-stand test | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. As physical parameters, the sit-to-stand test is performed (sec).
Correlation between protein-bound uremic toxin concentrations and muscle strength | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. Muscles strength is measured with handgrip test (N) and quadriceps test (N).
Correlation between protein-bound uremic toxin concentrations and risk of fall | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. An adaptation of the Dialysis Fall Risk Index is used as parameter for risk of fall (maximum score 12 - higher risk for higher score).
Correlation between protein-bound uremic toxin concentrations and nutritional status | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. Nutritional status is scored using the Mini Nutritional Assessment (MNA) questionnaire (score 24-30: normal nutritional status; 17-23.5: risk for malnutrition; 0-17: malnutrition)
Correlation between protein-bound uremic toxin concentrations and quality of life (EQ-5D) | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. Quality of life (QoL) is scored using the EQ-5D questionnaire (score 5-15 - lower QoL for higher score).
Correlation between protein-bound uremic toxin concentrations and quality of life (Promis) | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. Quality of life (QoL) is scored using the Promis questionnaire (standard deviation score - 40-60: normal score).
Correlation between protein-bound uremic toxin concentrations and objective sleep parameter (sleep efficiency) | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. The objective parameter 'sleep efficiency' (%) is derived from actigraphy measurement (better sleep for higher %).
Correlation between protein-bound uremic toxin concentrations and objective sleep parameter (fragmentation index) | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. The objective parameter 'fragmentation index' (higher score is worse) is derived from actigraphy measurement.
Correlation between protein-bound uremic toxin concentrations and patient survival | 10/2015 - 12/2018
  Blood samples are analysed for protein-bound toxins (mg/dL) in one High Performance Liquid Chromatography run. Survival is measured (in months).

OTHER OUTCOMES:
Difference between objectively measured sleep quality (sleep efficiency) in dialysis patients versus healthy controls | 2016-2018
  The objective parameter 'sleep efficiency' (%) is derived from actigraphy measurement and is compared between dialysis patients and age and gender matched healthy volunteers.
Difference between objectively measured sleep quality (fragmentation index) in dialysis patients versus healthy controls | 2016-2018
  The objective parameter 'fragmentation index' (higher score is worse) is derived from actigraphy measurement and is compared between dialysis patients and age and gender matched healthy volunteers.
Difference between subjectively measured sleep quality (ISI) in dialysis patients versus healthy controls | 2016-2018
  Subjective sleep parameter, as calculated from the Insomnia Severity Index (ISI) questionnaire, is compared between dialysis patients and age and gender matched healthy volunteers. The ISI score is 0-28 (the lower the better).
Difference between subjectively measured sleep quality (PSQI) in dialysis patients versus healthy controls | 2016-2018
  Subjective sleep parameter, as calculated from the Pittsburgh Sleep Quality Index (PSQI) questionnaire, is compared between dialysis patients and age and gender matched healthy volunteers. The ISI score is 0-27 (the lower the better).
Difference between the MNA scores for the short form (screening score) and the MNA score of the full form (indication score) | 10/2015-12/2018
  From the MNA questionnaire, the screening and indication scores are calculated and patients are for each score allocated to a group according to their score: i.e. normal nutritional status, risk for malnutrition, and malnutrition.
  Screening score: 12-14: normal nutritional status; 8-11: risk for malnutrition; 0-7: malnutrition.
  Indication score: 24-30: normal nutritional status; 17-23.5: risk for malnutrition; 0-17: malnutrition.
Correlation between subjective QoL score (EQ-5D) and physical parameter 6 minute walking test (6MWT) | 10/2015-12/2018
  Quality of life (QoL) is scored using the EQ-5D questionnaire (score 5-15). As physical parameters, the 6MWT (m) is performed.
Correlation between subjective QoL score (Promis) and physical parameter 6 minute walking test (6MWT) | 10/2015-12/2018
  Quality of life (QoL) is scored using the Promis questionnaire (standard deviation score).
  As physical parameters, the 6MWT (m) is performed.
Correlation between subjective QoL score (EQ-5D) and physical parameter sit-to-stand test | 10/2015-12/2018
  Quality of life (QoL) is scored using the EQ-5D questionnaire (score 5-15). As physical parameters, the sit-to-stand test (sec) is performed.
Correlation between subjective QoL score (Promis) and physical parameter sit-to-stand test | 10/2015-12/2018
  Quality of life (QoL) is scored using the Promis questionnaire (standard deviation score).
  As physical parameters, the sit-to-stand test (sec) is performed.
Correlation between subjective QoL score (EQ-5D) and muscle strength | 10/2015-12/2018
  Quality of life (QoL) is scored using the EQ-5D questionnaire (score 5-15). Muscle strength is measured with handgrip test (N) and quadriceps test (N).
Correlation between subjective QoL score (Promis) and muscle strength | 10/2015-12/2018
  Quality of life (QoL) is scored using the Promis questionnaire (standard deviation score).
  Muscles strength is measured with handgrip test (N) and quadriceps test (N).
Correlation between subjective QoL score (EQ-5D) and risk of fall | 10/2015-12/2018
  Quality of life (QoL) is scored using the EQ-5D questionnaire (score 5-15 - lower QoL for higher score).
  An adaptation of the Dialysis Fall Risk Index is used as parameter for risk of fall (maximum score 12 - higher risk for higher score).
Correlation between subjective QoL score (Promis) and risk of fall | 10/2015-12/2018
  Quality of life (QoL) is scored using the Promis questionnaire (standard deviation score - 40-60 normal score).
  An adaptation of the Dialysis Fall Risk Index is used as parameter for risk of fall (maximum score 12 - higher risk for higher score).
Correlation between subjective QoL score (EQ-5D) and nutritional status | 10/2015-12/2018
  Quality of life (QoL) is scored using the EQ-5D questionnaire (score 5-15). Nutritional status is scored using the Mini Nutritional Assessment (MNA) questionnaire (score 24-30: normal nutritional status; 17-23.5: risk for malnutrition; 0-17: malnutrition)
Correlation between subjective QoL score (Promis) and nutritional status | 10/2015-12/2018
  Quality of life (QoL) is scored using the Promis questionnaire (standard deviation score).
  Nutritional status is scored using the Mini Nutritional Assessment (MNA) questionnaire (score 24-30: normal nutritional status; 17-23.5: risk for malnutrition; 0-17: malnutrition)
Correlation between subjective QoL score (EQ-5D) and the objective sleep parameter (sleep efficiency) | 10/2015-12/2018
  Quality of life (QoL) is scored using the EQ-5D questionnaire (score 5-15). The objective parameter 'sleep efficiency' (%) is derived from actigraphy measurement.
Correlation between subjective QoL score (Promis) and the objective sleep parameter (sleep efficiency) | 10/2015-12/2018
  Quality of life (QoL) is scored using the Promis questionnaire (standard deviation score).
  The objective parameter 'sleep efficiency' (%) is derived from actigraphy measurement.
Correlation between subjective QoL score (EQ-5D) and the objective sleep parameter (fragmentation index) | 10/2015-12/2018
  Quality of life (QoL) is scored using the EQ-5D questionnaire (score 5-15). The objective parameter 'fragmentation index' (higher score is worse) is derived from actigraphy measurement.
Correlation between subjective QoL score (Promis) and the objective sleep parameter (fragmentation index) | 10/2015-12/2018
  Quality of life (QoL) is scored using the Promis questionnaire (standard deviation score).
  The objective parameter 'fragmentation index' (higher score is worse) is derived from actigraphy measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, PhD, MD, Principal Investigator — University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanden Wyngaert K, Celie B, Calders P, Eloot S, Holvoet E, Van Biesen W, Van Craenenbroeck AH. Markers of protein-energy wasting and physical performance in haemodialysis patients: A cross-sectional study. PLoS One. 2020 Jul 30;15(7):e0236816. doi: 10.1371/journal.pone.0236816. eCollection 2020. PMID 32730305